CLINICAL TRIAL: NCT03752944
Title: Stability of Maxillary Advancement by Lefort I Osteotomy in Patients With Retruded Maxilla Fixed With Two Prebent Plates Versus Four Miniplates. (Randomised Clinical Trial.)
Brief Title: Comparison Between Prebent & Miniplates in Fixation of Lefort I Osteotomty in Maxillary Advancement.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar Mahmoud Ahmed Mohamed, Resident of Oral and Maxillofacial Surgery - Nasser Institute Hospital for research & treatment / Master Candidate of Oral & Maxillofacial surgery, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-11-19
Record Dates: First submitted 2018-11-16; First posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Retruded Hypoplastic Maxilla

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant
Masking Description: Cards will have sequential numbers one number for each card then these cards will be placed within opaque sealed envelopes. Then these envelops will be placed in a container (box), each participant will grasp one envelope the day of procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prebent plate (Experimental): fixation of le fort I osteotomy using prebent plate
  Interventions: Procedure: lefort I osteotomy for maxillary advancement
- Conventional four miniplates (Active Comparator): fixation of le fort I osteotomy using conventional four miniplates
  Interventions: Procedure: lefort I osteotomy for maxillary advancement

INTERVENTIONS:
Procedure: lefort I osteotomy for maxillary advancement — fixation of lefort I osteotomy in patients with retruded maxilla with two prebent plates versus four miniplates.
  Other Names: four miniplates

SUMMARY:
In patients with retruded maxilla ,Will the use of two prebent plates produce more stable results postoperatively in fixation of Le Fort I osteotomy in maxillary advancement than conventional four minplates ? Many studies have been conducted to compare between the two plates and these studies showed that the prebent plate, the plate is not excessively twisted so that it can be adapted passively leading to less changes in the property of the material ,increased titanium contact surface to the bone leading to better force distribution resulting in better rigid fixation as no stresses will be transmitted from the plate to the bone leading to faster bone healing and consequently better long term postoperative stability.

DETAILED DESCRIPTION:
The stability of maxillary advancement after Le Fort I osteotomy in retruded maxilla patients has been an issue that has attracted the attention of numerous researchers. That's why different fixation methods have been compared in vitro and in vivo.

Prebent plates is one of the recent modifications of the plate systems used in maxillofacial surgery , they were created to reduce the need for bending and contouring of the titanium miniplates.

Lye et al.,(the only in vivo study in English), aimed to evaluate the predictability of advancement surgery with the use of prebent plates in 36 patients & he proved the prebent plates have been proven to significantly affect the advancement & reliable.

In a biomechanical study, prebent plates provided better results than the standard two plate scenario in terms of resistance to displacement, permanent deformation and load for breaking.

Fatih Mehmet Coskunses et al., in 2015 has done in vitro study to evaluate the segmental displacement, and von mises stress on the titanium miniplates & the maximum principal stress on the bone, with the use of prebent plates and two standard L plates adapted to either the zygomaticomaxillary buttress or the nasal piriform following anterior advancement of 5 mm or 10 mm by Le Fort I osteotomy.

The results of the study were, In 5 mm maxillary advancement using prebent plates for the fixation of bone segments resulted in less segmental displacement than the standard two plate.

Even when adapted posteriorly or anteriorly, the prebent plates were able to be more stable than two plates technique. Moreover, Not only the one prebent scenario had the lowest segmental displacements, but also the lowest maximum principal stresses on bone in the anteriorly adapted group.

These results are due to the structure of the prebent plates that have two arms extending in opposite directions (anteriorly and posteriorly) and it is suggested that the prebent plates are preferable alternatives to the traditional two plate configurations in osteotomies with up to 5 mm advancement. The prebent plates showed similar satisfactory results with 10 mm advancement only when adapted anteriorly. In contrast, when adapted posteriorly, the prebent plates resulted in obvious failure in the 10 mm advancement model.

Based on these data , My research will compare the postoperative stability between 2 groups of retruded maxilla patients having maxillary advancement up to 5 mm

1. the 1st group will be fixed using 2 prebent plates placed at nasal piriform
2. the 2nd group will be fixed using 4 miniplates placed at nasal piriform & zygmoaticomaxillay buttress.

The aim of this study:

To find out if the two prebent plates provides a stable postoperative maxillary advancement movement than the traditional four miniplates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with retruded maxilla & need advancement by le fort I osteotomy.
* Patients free from any systemic disease & bone metabolism diseases.
* Patients with no signs or symptoms of temporomandibular joint disorders.
* No sex predilection
* Age range ( 18-45)

Exclusion Criteria:

* Patients with systemic disease & bone metabolism diseases.
* Patients with cleft lip & palate.
* Patients with temporomandibular joint disorders
* Patients receiving chemotherapy or radiotherapy "due to the risk of low bone quality and healing
* Age less than 18

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Maxillary stability | 12 months
  Linear measurements (from A point to the nasion perpendicular, A point perpendicular to Frankfort plane) & Angular measurements (SNA , Maxillary depth angle ) will be obtained from the immediate postoperative lateral cephalometry and after 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hagar A Mohamed, BDS, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coskunses FM, Kan B, Mutlu I, Cilasun U, Celik T. Evaluation of prebent miniplates in fixation of Le Fort I advancement osteotomy with the finite element method. J Craniomaxillofac Surg. 2015 Oct;43(8):1505-10. doi: 10.1016/j.jcms.2015.07.004. Epub 2015 Jul 15. PMID 26297421